CLINICAL TRIAL: NCT00881062
Title: A Phase 1 Study to Investigate the Absorption, Metabolism and Excretion of [14C}-Proellex Following Single Oral Dose Administration in Healthy Female Subjects
Brief Title: Investigate Absorption, Metabolism and Excretion of [14C}-Proellex Following Single Oral Dose in Healthy Females
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Repros Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: ZP-009
Record Dates: First submitted 2009-04-14; First posted 2009-04-15 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: ABSORPTION; METABOLISM; EXCRETION
Keywords: ABSORPTION; METABOLISM; EXCRETION
MeSH Terms: interventions — telapristone acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 25 mg Proellex (Experimental): 25 mg (100 µCi) [14C]-Proellex
  Interventions: Drug: Proellex

INTERVENTIONS:
Drug: Proellex — A single oral dose administered after at least a 10 hour fast
  Other Names: Telapristone acetate

SUMMARY:
This study was to determine the ADME and metabolites of Proellex following a single oral dose of 25 mg.

DETAILED DESCRIPTION:
The purpose of this study is to determine the absorption, metabolism, and excretion kinetics of Proellex and to determine and characterize metabolites present in plasma and urine following a single oral dose of 25 mg. The 25 mg dose selected for this study has been included in all previous clinical trials. This dose was well tolerated and demonstrated efficacy against uterine fibroids and endometriosis.

ELIGIBILITY:
Inclusion Criteria:

* In good health, determined by no clinically significant findings from medical history, 12-lead ECG, and vital signs
* Clinical laboratory evaluations within the reference range for the test laboratory, unless deemed not clinically significant by the Investigator
* 1 to 2 bowel movements per day.

Exclusion Criteria:

* Significant history or significant clinical manifestation (as determined by the Investigator) of any metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, or psychiatric disorder
* History of stomach or intestinal surgery or resection that would potentially alter absorption and/or excretion of orally administered drugs
* Participation in more than 1 other radiolabeled investigational study drug trial within 12 months prior to check-in
* Exposure to significant radiation (eg, serial x-ray or computed tomography scans, barium meal, current employment in a job requiring radiation exposure monitoring) within 12 months prior to check-in
* Donation of blood from 30 days prior to Screening through Clinic Discharge, inclusive, or of plasma from 2 weeks prior to Screening through clinic discharge, inclusive
* Receipt of blood products within 2 months prior to check-in

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2009-04; Primary Completion 2009-05 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
To assess the pharmacokinetics (PK) of a single dose of Proellex and its metabolites using [14C]-Proellex | 14 days

SECONDARY OUTCOMES:
To characterize and identify metabolites of [14C]-Proellex in plasma and urine | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Andre van As, MD, PhD, Study Director — Repros Therapeutics Inc.
Locations (1):
- Covance Clinical Research Unit Inc., Madison, Wisconsin, United States